CLINICAL TRIAL: NCT00182507
Title: A 12-Week, Double-Blind Trial of Olanzapine and Placebo in the Treatment of Trichotillomania
Brief Title: Olanzapine in the Treatment of Hair Pulling (Trichotillomania)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Eli Lilly and Company (Industry)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-167
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-03

CONDITIONS: Trichotillomania
MeSH Terms: conditions — Trichotillomania | interventions — Olanzapine

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
Trichotillomania (TTM) or hair-pulling has been considered as part of the obsessive compulsive disorder (OCD) spectrum, although treatment with OCD medications has largely been unsuccessful. Tics/Tourrettes' Syndrome (TS) is a disorder, which appears to be related to TTM, but is treated with a different class of medications than used in OCD, namely antipsychotics such as olanzapine. This is a study of the safety and efficacy of olanzapine in the treatment of hair pulling.

ELIGIBILITY:
Inclusion Criteria:

* primary DSM-IV trichotillomania; CGI-Severity ≥ 4

Exclusion Criteria:

* Any other Axis I primary diagnosis; CGI-S < 4; current comorbid: OCD, MDD, alcohol or substance abuse; lifetime hx of: schizophrenia, bipolar affective disorder or dementia; current pregnancy/lactation; current suicidality or homicidality; major medical problems or clinically unstable medical disease; hx of: seizures, stroke or head trauma; prior use of neuroleptics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2000-06; Study Completion 2006-03

PRIMARY OUTCOMES:
Clinical Global Impression (CGI)-Improvement Scale ≤ 2

SECONDARY OUTCOMES:
CGI-Severity Scale, Mean change from baseline in: Yale-Brown Obsessive Compulsive Scale for TTM, the Massachusetts General Hospital Hair Pulling Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Van Ameringen, MD, FRCPC, Principal Investigator — Hamilton Health Science, McMaster Univeristy Medical Centre
Locations (1):
- Hamilton Health Sciences, McMaster University Medical Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562
- [Derived] Van Ameringen M, Mancini C, Patterson B, Bennett M, Oakman J. A randomized, double-blind, placebo-controlled trial of olanzapine in the treatment of trichotillomania. J Clin Psychiatry. 2010 Oct;71(10):1336-43. doi: 10.4088/JCP.09m05114gre. Epub 2010 Apr 20. PMID 20441724